CLINICAL TRIAL: NCT00280267
Title: Testosterone Therapy After Hip Fracture in Elderly Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Ellen Binder, MD, Washington University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R21AG023716 (NIH)
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Hip Fracture; Testosterone Deficiency; Muscle Weakness
Keywords: hip fracture; testosterone; muscle weakness; frail elderly; aging
MeSH Terms: conditions — Hip Fractures; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Testosterone gel

SUMMARY:
The purpose of this study is to determine the feasibility of testosterone replacement therapy in frail elderly female hip fracture patients who have testosterone deficiency, and to obtain preliminary information about the effects of testosterone therapy on muscle strength and size, bone density, mobility, daily functioning, and quality of life.

DETAILED DESCRIPTION:
Hip fractures are common among elderly women and can have a devastating impact on their ability to remain independent. A significant functional decline following a hip fracture has been documented, and many patients have persistent strength and mobility deficits that impair their capacity for independent function. Such individuals are at high risk for continued supportive services, recurrent injury, and institutionalization. High-risk patients include those with deficits in skeletal muscle strength during the post-fracture period. Age-associated androgen deficiency contributes to deficits in muscle mass and strength that are common in this patient population. The role of testosterone therapy for improving deficits in muscle mass, strength, and functional capacity in the frail elderly is unclear, particularly for elderly women. There is insufficient information regarding tolerability of testosterone therapy, and the appropriate medication dosage and target serum testosterone levels necessary to induces changes in skeletal muscle mass and functional measures in elderly women with physical frailty due to muscle weakness.

The goals of this project are to conduct a randomized, double-blinded, placebo-controlled prospective study to determine the feasibility, tolerability, and safety of 6 months of testosterone therapy in community-dwelling, physically frail, elderly female hip fracture patients. Twenty-seven female hip fracture patients will be recruited, using objective criteria for testosterone deficiency and frailty. We plan to evaluate two dosages of testosterone, administered as a 0.5% topical gel: a physiologic replacement dosage, and a supraphysiologic dosage. We plan to carefully monitor testosterone levels, side effects, biochemical parameters, and factors related to compliance with therapy. We plan to obtain preliminary information regarding the changes in measurements of muscle strength, total score on an Objective Physical Performance Test, total lean body mass by dual energy x-ray absorptiometry (DEXA), thigh cross-sectional areas by magnetic resonance imaging (MRI), and self-reported performance of activities of daily living, and quality of life. These data will be used to develop a full-scale proposal to test the long-term hypothesis that testosterone therapy combined with exercise training can improve physical function after a hip fracture.

ELIGIBILITY:
Inclusion Criteria: -female, hip fracture repair within previous 4 months

* age 65 years and older
* serum total testosterone level < 30 ng/dl
* modified Physical Performance Test Score between 13-28
* able to ambulate 50 ft

Exclusion Criteria: -permanent nursing home residence

* dementia severe enough to prohibit informed consent
* clinically significant visual or hearing impairments
* history of a hormone dependent neoplasia
* active or unstable cardiopulmonary disease
* history of sleep apnea
* elevated liver function tests
* hematocrit > 51%
* history of alcohol or substance abuse
* symptoms of depression severe enough to cause weight loss of >5% in previous 3 months or interfere with daily activities or medication compliance

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Serum testosterone levels, drug compliance, symptoms and side effects during the six months of treatment. | Six months

SECONDARY OUTCOMES:
Modified Physical Performance Test Score at 6 months | Six months
1-RM muscle strength at 6 months | Six months
Thigh cross-sectional area by MRI at 6 months | Six months
Self-report of ADL function at 6 months | Six months
SF-36 score (quality of life) at 6 months | Six months
Total and regional bone density by DEXA at 6 months | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F. Binder, MD, Principal Investigator — Washington University School of Medicine, Division of Geriatrics and Nutritional Science
Locations (1):
- Washington University School of Medicine, Division of Geriatrics and Nutritional Science, St Louis, Missouri, United States